CLINICAL TRIAL: NCT02094638
Title: Post-Marketing Surveillance of the Tanreqing Injection: a Real World Study
Status: Completed | Type: Observational
Sponsor: Suodi ZHAI (Other)
Collaborators: Shanghai Kaibao Pharmaceutical CO.,LTD. (Unknown); Peking University (Other); Handan First Hospital (Other); Bethune International Peace Hospital of the Chinese PLA (Unknown); The 254th Hospital of chinese People's Liberation Army (Unknown); The 464th Hospital of chinese People's Liberation Army (Unknown); People's Hospital of Cangzhou (Unknown); The First Hospital of Qinhuangdao (Other Government); The 44th Hospital of chinese People's Liberation Army (Unknown); First Affiliated Hospital of Kunming Medical University (Other); The Second Affiliated Hospital of Kunming Medical University (Other); Chongqing Three Gorges Central Hospital (Other); Sichuan Provincial People's Hospital (Other); ShuangLiu Hospital of Traditional Chinese Medical (Unknown); People's Hospital of Nanbu County (Unknown); DuJiangyan Traditional Chinese Medicine Hospital (Unknown); West China Hospital (Other); Chongqing Traditional Chinese Medicine Hospital (Other); The Third People's Hospital of Chongqing (Unknown); Changsha Fourth Hospital (Other Government); Hubei Xinhua Hospital (Other); Wenzhou Central Hospital (Other); Affiliated Yueqing Hospital of Wenzhou Medical University (Other); The First Affiliated Hospital of Nanchang University (Other); Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other); Shanghai Minhang District Central Hospital (Unknown); Shanghai First People's Hospital Branch (Unknown); Zhejiang Provincial Hospital of TCM (Other); The Affiliated Hospital of Hainan medical College (Unknown); Guiyang Children's Hospital (Unknown); Traditional Chinese Medical Hospital of Jiangxi Province (Unknown); Jiangxi Provincial People's Hopital (Other); Hubei Cancer Hospital (Other); Jiangning District Hospital of Traditional Chinese Medicine (Unknown); Shenzhen Third People's Hospital (Other); Ningbo No. 1 Hospital (Other); Second Hospital of Jilin University (Other); The First Hospital of Jilin University (Other); Yangzhou No.1 People's Hospital (Other); Traditional Chinese Medical Hospital of Bai Autonomous Prefecture of Dali (Unknown); Bijie First Municipal People's Hospital (Unknown); Guiyang Pulmonary Hospital (Unknown); The 263rd Hospital of Chinese People's Liberation Army (Unknown); Chongqing Kaixian County People's Hospital (Unknown); The Second Affiliated Hospital of Chongqing Medical University (Other); Chongqing Jiulongpo First People's Hospital (Unknown); People's Hospital of Xinjiang Uygur Autonomous Region (Other); Shenyang 242 Hospital (Unknown); Second Affiliated Hospital of Guangzhou Medical University (Other); Cancer Hospital of Guizhou Province (Other); Wu Song Central Hospital of Shanghai (Unknown); Gansu Provincial Hospital (Other); Lanzhou Petrochemical General Hospital (Unknown); Traditional Chinese Medicine Hospital of the Ningxia Hui Autonomous Region (Other); General Hospital of Ningxia Medical University (Other); The First People's Hospital of Yinchuan (Other); Yantai Municipal Laiyang Central Hospital (Unknown); Shandong Cancer Hospital and Institute (Other); Shandong University of Traditional Chinese Medicine (Other); Zunyi Medical College (Other); The 152nd Hospital of chinese People's Liberation Army (Unknown); Henan Provincial People's Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Central South University (Other); The Second Hospital of Nanchang (Unknown); The Second Hospital of Wulanchabu City (Unknown); Qinghai Women and Childhood Hospital (Unknown); The Third People's Hospital of Chengdu (Other); The Center Hospital of Shuozhou (Unknown); Yunnan Provinical Hospital of Traditional Chinese Medicine (Other); Beijing Geriatric Hospital (Other); Hubei Zhongshan Hospital Affiliated to Wuhan University (Unknown); Anhui Provincial Children's Hospital (Other); The Third Affiliated Hospital of Inner Mongolia Medical College (Unknown); The fourth Hospital of Inner Mongolia (Unknown); Zhongshan People's Hospital, Guangdong, China (Other); Fenyang Hospital of Shanxi Province (Unknown); The First Hospital Of Huhhot (Unknown); Taiyuan Xinghualing Maternity & Child Health Care Center (Other); The Fifth People's Hospital of Datong (Unknown); Shanxi Provincial Maternity and Children's Hospital (Other); The Second People's Hospital of Jinzhong (Unknown); The Second Hospital of Hebei Medical University (Other); People's Hospital of Rongcheng (Unknown); Hebei Zhaoxian People's Hospital (Unknown); Hejian Municipal People's Hospital (Unknown); Xinle Municipal Hospital of Hebei (Unknown); Capital Medical University (Other); Fengtai district Hospital of Chinese and Western medicine, Beijing (Unknown); Shanghai Changzheng Hospital (Other); Xintai People's Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Suodi ZHAI, Suodi ZHAI, Department of Pharmacy, Peking University Third Hospital, Peking University Third Hospital
Organization: Peking University Third Hospital (Other)
Other Study IDs: PekingUTH-Pharmacy-003
Record Dates: First submitted 2014-03-20; First posted 2014-03-24 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Adverse Drug Reaction; Drug Allergy
Keywords: Traditional Chinese Medicine Injection
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Drug Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Biospecimen Retention: Samples With DNA — biospecimen including serum, plasma, blood cells with DNA.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Tanreqing: Inpatient using the Tanreqing Injection

SUMMARY:
Tanreqing Injection is widely used in respiratory disease with Chinese medicine syndrome of retention of phlegm and heat in Fei. This study record clinical use of Tanreqing Injection in the real world, observe the adverse drug reactions/ adverse drug events during treatment, and figure out why Tanreqing induced severe allergic reaction happens.

DETAILED DESCRIPTION:
As a compound traditional Chinese medicine, Tanreqing Injection was approved by China Food and Drug Administration(CFDA) in 2003, and widely used respiratory disease, such as biofilm related upper respiratory infections, pneumonia and bronchitis. During its 11 years marketing in China, there was hardly any serious adverse drug reactions except for a few cases reported as severe allergic reaction. In this study, clinical pharmacists in selected hospitals will not only record the clinical use and the adverse drug reactions/ adverse drug events of this injection, but also try to figure out why drug-induced severe allergic reaction happens through a nested case-control study. This real world study for Tanreqing Injection with 30400 patients will be conducted from January.2014 to June.2016.

ELIGIBILITY:
Inclusion Criteria:

* Patients who use the Tanreqing Injection in selected hospitals in China, including inpatient and outpatient.
* Outpatients will be only in some hospitals which can get the patients' complete information.

Exclusion Criteria:

* Patients who are less than 24 months.

Min Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who use the Tanreqing Injection in selected hospitals in China (including the inpatient and the outpatient(only in some hospitals which can get the information)).
Sampling Method: Non-Probability Sample
Enrollment: 30400 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse drug reaction of Tanreqing Injection | 30 months

SECONDARY OUTCOMES:
Outcomes of the patients who experienced an adverse drug reaction of Tanreqing Injection | 30 months
  Outcomes including cure, improved, null, or death.
Administration of Tanreqing Injection in real world | 30 months
Population characteristics of the adverse drug reaction of Tanreqing Injection | 30 months
Off-lable use of Tanreqing Injection | 30 months
Drug combination of Tanreqing Injection in real world | 30 months

OTHER OUTCOMES:
Related Risk Factors in severe allergic reaction of Tanreqing Injection | 30 months

CONTACTS AND LOCATIONS:
Locations (90):
- China (90):
  - Anhui Provincial Children's Hospital, Hefei, Anhui
  - The Fengtai district Hospital of Integrated TCM & WM, Beijing, Beijing Municipality
  - Beijing Geriatric Hospital, Beijing, Beijing Municipality
  - The 263rd Hospital of Chinese People's Liberation Army, Beijing, Beijing Municipality
  - Beijing Luhe Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The Third People's Hospital of Chongqing, Chongqing, Chongqing Municipality
  - Chongqing Traditional Chinese Medicine Hospital, Chongqing, Chongqing Municipality
  - Chongqing Jiulongpo First People's Hospital, Chongqing, Chongqing Municipality
  - Chongqing Three Gorges Central Hospital, Chongqing, Chongqing Municipality
  - Chongqing Kaixian County People's Hospital, Chongqing, Chongqing Municipality
  - Gansu Provincial Hospital of Traditional Chinese Medicine, Lanzhou, Gansu
  - Lanzhou Petrochemical General Hospital, Lanzhou, Gansu
  - The Third People's Hospital of Huizhou, Huizhou, Guangdong
  - The Third People's Hospital of Shenzhen, Shenzhen, Guangdong
  - Zhongshan Municipal People's Hospital, Zhongshan, Guangdong
  - Bijie First Municipal People's Hospital, Bijie, Guizhou
  - Guiyang Children's Hospital, Guiyang, Guizhou
  - Guiyang Pulmonary Hospital, Guiyang, Guizhou
  - Guizhou Cancer Hospital, Guiyang, Guizhou
  - The 44th Hospital of chinese People's Liberation Army, Guiyang, Guizhou
  - Affiliated Hospital of Zunyi Medical College, Zunyi, Guizhou
  - The Affiliated Hospital of Hainan medical College, Haikou, Hainan
  - People's Hospital of Rongcheng, Baoding, Hebei
  - People's Hospital of Cangzhou, Cangzhou, Hebei
  - First Hospital of Handan City, Handan, Hebei
  - Hejian Municipal People's Hospital, Hejian, Hebei
  - The First Hospital of Qinhuangdao, Qinhuangdao, Hebei
  - the Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Bethune International Peace Hospital of the Chinese PLA, Shijiazhuang, Hebei
  - Hebei Zhaoxian People's Hospital, Shijiazhuang, Hebei
  - Xinle Municipal Hospital of Hebei, Xinle, Hebei
  - The 152nd Hospital of chinese People's Liberation Army, Pingdingshan, Henan
  - Henan Province Hospital of TCM, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hubei Xinhua Hospital, Wuhan, Hubei
  - Hubei Zhongshan Hospital Affiliated to Wuhan University, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - The Fourth Hospital of Changsha, Changsha, Hunan
  - the Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The Third Affiliated Hospital of Inner Mongolia Medical College, Baotou, Inner Mongolia
  - The First Hospital Of Huhhot, Hohhot, Inner Mongolia
  - The fourth Hospital of Inner Mongolia, Hohhot, Inner Mongolia
  - The Second Hospital of Wulanchabu City, Wulanchabu, Inner Mongolia
  - Jiangning District Hospital of Traditional Chinese Medicine, Nanjing, Jiangsu
  - The First People's Hospital of Yangzhou City, Yangzhou, Jiangsu
  - The Second Hospital of Nanchang, Nanchang, Jiangxi
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - Traditional Chinese Medical Hospital of Jiangxi Province, Nanchang, Jiangxi
  - The First Hospital of Nanchang, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - The Second Hospital of Jilin University, Changchun, Jilin
  - Shenyang 242 Hospital, Shenyang, Liaoning
  - The First People's Hospital of Yinchuan, Yinchuan, Ningxia
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Chinese Traditional Medicine Hospital of Ningxia Autonomous Region, Yinchuan, Ningxia
  - Qinghai Women and Childhood Hospital, Xining, Qinghai
  - Affiliated Hospital of Shandong University of Traditional Chinese Medicine, Jinan, Shandong
  - Shandong Cancer Hospital, Jinan, Shandong
  - Xintai People's Hospital, Xintai, Shandong
  - Yantai Municipal Laiyang Central Hospital, Yantai, Shandong
  - Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality
  - Shanghai Ninth People's Hospital, Shanghai JiaoTong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai First People's Hospital Branch, Shanghai, Shanghai Municipality
  - Wu Song Central Hospital of Shanghai, Shanghai, Shanghai Municipality
  - Shanghai Minhang District Central Hospital, Shanghai, Shanghai Municipality
  - Fifth Hospital of Datong, Datong, Shanxi
  - Fenyang Hospital of Shanxi Province, Fenyang, Shanxi
  - The Second People's Hospital of Jinzhong, Jinzhong, Shanxi
  - The Center Hospital of Shuozhou, Shuozhou, Shanxi
  - Maternal and Child Health Care Hospital of Taiyuan, Taiyuan, Shanxi
  - Shanxi Maternity and Children Health Hospital, Taiyuan, Shanxi
  - The Third People's Hospital of Chengdu, Chengdu, Sichuan
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - ShuangLiu Hospital of Traditional Chinese Medical, Chengdu, Sichuan
  - DuJiangyan Traditional Chinese Medicine Hospital, Dujiangyan, Sichuan
  - People's Hospital of Nanbu County, Nanchong, Sichuan
  - The 254th Hospital of chinese People's Liberation Army, Tianjin, Tianjin Municipality
  - The 464th Hospital of chinese People's Liberation Army, Tianjin, Tianjin Municipality
  - People's Hospital of Xinjiang Uigur Autonomous Region, Ürümqi, Xinjiang
  - Traditional Chinese Medical Hospital of Bai Autonomous Prefecture of Dali, Dali, Yunnan
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Zhejiang Provincial Hospital of TCM, Hangzhou, Zhejiang
  - Ningbo First Hospital, Ningbo, Zhejiang
  - Wenzhou Central Hospital, Wenzhou, Zhejiang
  - The Second Affiliated Hospital of Wenzhou Medical College, Wenzhou, Zhejiang
  - Wenzhou Yueqing People's Hospital, Wenzhou, Zhejiang
  - Peking university third hospital, Beijing